CLINICAL TRIAL: NCT04996641
Title: A Clinical Trial Pilot Study Investigating a New Dental Protocol for Pre-Radiation Endodontic-Restorative Therapy of Head and Neck Cancer Patients
Brief Title: Endodontic-Restorative Pre-Radiation Therapy of Head and Neck Cancer Patients
Acronym: EndoRest
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll participants
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: University of Zagreb (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 06321
Record Dates: First submitted 2021-05-21; First posted 2021-08-09 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2022-03

CONDITIONS: Pulpitis - Irreversible; Caries; Head and Neck Cancer
Keywords: Restoration; Tooth Retention
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Crowns

STUDY DESIGN:
Intervention Model Description: This study involves a modified, expedited tooth restoration procedure for individuals scheduled to undergo radiation therapy for head and neck cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Root canal treatment and crown restoration
  Interventions: Procedure: Root canal treatment and crown

INTERVENTIONS:
Procedure: Root canal treatment and crown — Pre-radiation one day root canal treatment and CAD/CAM chair side fabricated crowns for head and neck cancer patients

SUMMARY:
Pilot study involving 20 patients undergoing dental treatment prior to radiation therapy. Comparison of outcome parameters to existing data of age and gender matched patients.

DETAILED DESCRIPTION:
Advanced radiation therapy systems are part of head/neck cancer treatment. 2-3 weeks prior to the initiation of radiation therapy (preRT), patients undergo dental screening, simple restorations and the removal of teeth deemed a osteoradionecrosis risk, often including asymptomatic, vital teeth. Time limitations preRT generally prohibit a traditional multi-visit approach for endodontic treatment, crown preparation, and an externally fabricated restoration. Precision restorative dentistry, with CAD/CAM milled ceramic restorations allow for immediate post-endodontic rehabilitation on the same. The Center for Clinical and Translational Research (CCTR) at PDM conducts the ARMOR trial, a randomized, controlled trial testing the efficacy of two oral care protocols enrolling 120 cancer patients from the Perelman Center for Advanced Medicine (PCAM) over 3.5 years. This pilot study will enroll 20 patients of the ARMOR trial for endodontic treatment and restoration of posterior asymptomatic and vital teeth using microscopic endodontics and digital precision CAD/CAM restoration. These teeth would otherwise be extracted due to time limitations preRT. Patients will be seen for the dental treatment within the time window from diagnosis to initiation of radiation therapy. Patients will be evaluated for (1) feasibility of the suggested protocol (primary objective); quality of life as in the ARMOR trial; 2) tooth survival; 3) endodontic status [PAI index]; 4) periodontal prognosis and status [McGuire-Nunn Criteria, etc]; and 5) restorative status [USPHS Criteria, etc] (secondary objectives) at 1,2,5 months follow-ups of the ARMOR trial. For control, data for tooth survival and QLQ will be compared to 20 other participants of the ARMOR trial (10/10 per study arm) that do not participate in the EndoRest substudy and to 20 other matching participants patients (age, gender) from an existing, comparable dataset of the ORA-RAD studies of the Penn Study arm at PDM Oral Medicine. Periodontal status and restorative status (iff applicable) will be compared to contra-lateral or counter-arch teeth of the individual participant.

ELIGIBILITY:
Inclusion Criteria:

1. Patient volunteering to participate in the study.
2. Patients eligible for participation in the ARMOR trial (current head and neck cancer patient trial conducted at Penn Dental Medicine[PDM])
3. Non-contributory medical history (Patient can be seen for dental appointment in PDM).
4. No history of previous endodontic treatment on the tooth/teeth selected for treatment.
5. Asymptomatic and vital teeth with deep decay (Irreversible pulpitis due to decay reaching pulp).

Exclusion Criteria:

Economic status, gender, race or ethnicity are not of concern for the proposed investigation and therefore for study exclusion. Patients will not be eligible to participate in the study if any of the following exclusion criteria applies:

1. Symptoms or necrotic tooth with presence of periapical radioluceny.
2. History of previous endodontic treatment on the teeth to be treated.
3. Teeth affected by fractures.
4. Compromised periodontal status with pockets exceeding 4 mm, exceeding mobility I or gingival edema).
5. At the discretion of the PI, patient is unlikely or unwilling to follow study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with successful completion of endodontic and restorative treatment of teeth (Feasibility) | 1-5 days
  Evaluation of whether the proposed one-day root canal treatment plus crown restoration protocol can be utilized and executed prior to radiation treatment of head and neck cancer patients. The evaluation will be on a per patient, not per tooth, basis. Failure is defined as the inability to complete endodontic treatment and definitive restoration of a qualifying tooth in a study participant, resulting in the need for pre-radiation extraction of the tooth.
Delay in RT initiation, calculated on a scale of 0-100 for the study, as described below (Feasibility) | 2-10 days
  Evaluation of whether the onset of radiation therapy was delayed due to participation in the EndoRest study. The evaluation will be on a per patient, not per tooth, basis. Delay in RT start will be scored on the following scale:
  5 points: RT started as planned; no delays 4 points: RT delayed by 1 day due to participation in the EndoRest study 3 points: RT delayed by 2 days due to participation in the EndoRest study 2 points: RT delayed by 3 days due to participation in the EndoRest study 0 points: RT delated by 4 or more days due to participation in the EndoRest study
  The total points for all participants in the study will be summed. A score of >=90 indicated that the protocol is feasible. A total score <90 indicates that the protocol is not feasible.
Number of participants who need post-radiation extraction of a qualifying tooth. | 5 months
  Evaluation of whether a qualifying tooth for which endodontic and restorative treatment was successfully completed was extracted in the time interval post-radiation therapy up to 5 months after the initial visit.

SECONDARY OUTCOMES:
Evaluation of quality of life (QOL) based on the EORTC-QLQ-C30 | 5 months
  Quality of life and function will be assessed using the validated European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) with the Head and Neck specific questionnaire add-on (HN43). This questionnaire assesses general quality of life as well as issues specific to head and neck cancer patients (e.g. difficulty swallowing, pain, dry mouth).
  All questions on the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire EORTC-QLQ are assigned a score of 0-100. A higher score indicates a higher response level (for function questions, a high score indicates a high level of function, indicating a better outcome. For symptom questions, a high score indicates a high level of symptomology, indicating a worse outcome).
Evaluation of tooth survival | 5 months
  Tooth survival after completion of endodontic-restorative treatment will be assessed in all participants using standard survival analysis techniques.
Evaluation of endodontic status using the PAI | 5 months
  Endodontic status will be assessed using the periapical index (PAI). PAI uses a scale of 0-5, with 0 meaning "healthy" and 5 meaning "severe periodontitis with exacerbated features."
Evaluation of periodontal status | 5 months
  Periodontal status will be assessed through probing depths of periodontal pockets of the treated tooth.
Evaluation of restorative status using the USPHS criteria | 5 months
  Restoration status will be assessed using United States Public Health System (USPHS) criteria. The USPHS criteria assesses anatomical form, marginal adaptation, color match, marginal discoloration, surface roughness, and caries, in a single assessment tool. Higher scores indicate less favorable outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Setzer, DMD, PhD, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- School of Dental Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be made available to other researchers.

REFERENCES:
- [Background] Kataoka SH, Setzer FC, Fregnani ER, Pessoa OF, Gondim E Jr, Caldeira CL. Effects of 3-dimensional conformal or intensity-modulated radiotherapy on dental pulp sensitivity during and after the treatment of oral or oropharyngeal malignancies. J Endod. 2012 Feb;38(2):148-52. doi: 10.1016/j.joen.2011.09.022. Epub 2011 Nov 14. PMID 22244627
- [Background] Kataoka SH, Setzer FC, Gondim-Junior E, Fregnani ER, Moraes CJ, Pessoa OF, Gavini G, Caldeira CL. Late Effects of Head and Neck Radiotherapy on Pulp Vitality Assessed by Pulse Oximetry. J Endod. 2016 Jun;42(6):886-9. doi: 10.1016/j.joen.2016.02.016. Epub 2016 Apr 9. PMID 27071975
- [Background] Wahl MJ. Osteoradionecrosis prevention myths. Int J Radiat Oncol Biol Phys. 2006 Mar 1;64(3):661-9. doi: 10.1016/j.ijrobp.2005.10.021. PMID 16458773
- [Background] Nabil S, Samman N. Incidence and prevention of osteoradionecrosis after dental extraction in irradiated patients: a systematic review. Int J Oral Maxillofac Surg. 2011 Mar;40(3):229-43. doi: 10.1016/j.ijom.2010.10.005. Epub 2010 Nov 5. PMID 21115324
- [Background] Chang DT, Sandow PR, Morris CG, Hollander R, Scarborough L, Amdur RJ, Mendenhall WM. Do pre-irradiation dental extractions reduce the risk of osteoradionecrosis of the mandible? Head Neck. 2007 Jun;29(6):528-36. doi: 10.1002/hed.20538. PMID 17230555
- [Background] Ben-David MA, Diamante M, Radawski JD, Vineberg KA, Stroup C, Murdoch-Kinch CA, Zwetchkenbaum SR, Eisbruch A. Lack of osteoradionecrosis of the mandible after intensity-modulated radiotherapy for head and neck cancer: likely contributions of both dental care and improved dose distributions. Int J Radiat Oncol Biol Phys. 2007 Jun 1;68(2):396-402. doi: 10.1016/j.ijrobp.2006.11.059. Epub 2007 Feb 22. PMID 17321069
- [Background] Clayman L. Clinical controversies in oral and maxillofacial surgery: Part two. Management of dental extractions in irradiated jaws: a protocol without hyperbaric oxygen therapy. J Oral Maxillofac Surg. 1997 Mar;55(3):275-81. doi: 10.1016/s0278-2391(97)90542-5. No abstract available. PMID 9054917
- [Background] Hentz C, Diaz AZ, Borrowdale RW, Emami B, Kase M, Choi M. Establishing a targeted plan for prophylactic dental extractions in patients with laryngeal cancer receiving adjuvant radiotherapy. Oral Surg Oral Med Oral Pathol Oral Radiol. 2016 Jul;122(1):43-9. doi: 10.1016/j.oooo.2016.01.021. Epub 2016 Feb 13. PMID 27068679